CLINICAL TRIAL: NCT02136160
Title: Rakuns: Setting-based Prevention Program to Promote Positive Experiences in Health Promoting Lifestyle Choices
Brief Title: Population-based Intervention to Promote Health in Elementary Schools
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: Child Health Foundation (Other); Johnson & Johnson Citizenship Trust, in cooperation with Johnson & Johnson GmbHInitiative Rückenwirbel e.V., Gmund (Unknown); Platform for Diet and Physical activity e.V. (peb) (Unknown)
Responsible Party: Principal Investigator, Prof. Berthold Koletzko, Berthold Koletzko, M.D., Professor of Paediatrics, Dr. von Hauner Children´s Hospital, Ludwig-Maximilians-University, Munich, Germany, Ludwig-Maximilians - University of Munich
Allocation: Not Applicable | Masking: None | Purpose: Prevention
Other Study IDs: Rakuns
Record Dates: First submitted 2014-05-05; First posted 2014-05-12 (Estimated); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Health Promotion
Keywords: elementary school; children; health promotion; teachers; prevention
MeSH Terms: interventions — National Program of Cancer Registries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: attitude change, behavioral change
Behavioral: prevention program

SUMMARY:
Population based intervention at elementary school setting aimed at contributing, to a major extent, to health education and health promotion for children aged approximately 5-10 years in Germany. Health education units with theoretical and practical exercises for use by teachers, children, and parents addresses physical activity, sedentary behavior, relaxation, nutrition, personal hygiene and body awareness.

Main questions of the pilot are:

Does health promotion take on an important role in primary schools? How do teachers evaluate training materials, homepage, content and framework conditions? How do teachers assess the efficiency of teaching units?

DETAILED DESCRIPTION:
The program is based on actual cognitions and methods of the early education science. In the pilot phase study part (3/2013-5/2013) the investigators evaluated 210 classes of five states in Germany: NRW, Thüringen, Berlin, Sachsen-Anhalt, Schleswig-Holstein.

The long-term aim of this project is to provide an innovative concept based on current concepts in social studies and science that addresses health education of pupils in elementary schools.

ELIGIBILITY:
Inclusion Criteria:

* teacher of intervention-school

Exclusion Criteria:

* absence of consent to participate

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Start 2013-03; Primary Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Change of health related behaviour due to intervention | After 6 weeks of intervention period

REFERENCES:
- See also: project website — http://rakuns.de